CLINICAL TRIAL: NCT06928883
Title: TITAN-PARADISE Pilot: TicIn for the Treatment of Coronary Lesions - Plaque Regression and Stabilization With Sirolimus Elution (Pilot Study)
Brief Title: Ticin Pilot Study: Sirolimus-Eluting Balloon for Stabilization and Regression of Non-Obstructive Coronary Plaques.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cardiocentro Ticino (Other)
Responsible Party: Principal Investigator, Marco Valgimigli, Prof. Dr. Med. Marco Valgimigli, Deputy Chief, Cardiocentro Ticino
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TITAN-PARADISE Pilot
Record Dates: First submitted 2025-03-11; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Coronary Arterial Disease (CAD); Vulnerable Coronary Plaques; Multivessel Coronary Artery Disease; Coronary Vessel; Acute Coronary Syndromes (ACS)
Keywords: Coronary Arterial Disease (CAD); Vulnerable Coronary Plaques; Multivessel coronary artery disease; Coronary vessel; Acute Coronary Syndromes (ACS); Non-flow limiting vulnerable coronary plaques; Sirolimus-eluting DEB; DEB Selution SLR; Guidelines-directed medical therapies (GDMT); IVUS-NIRS; MaxLCBI4mm; MaxLCBI4mm≥325; Lipid Core Burden Index (LCBI)
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sirolimus-eluting DEB (Selution SLR) therapy + Guidelines-directed medical therapy (Experimental): Selution SLR sirolimus-eluting balloon additional to guidelines-directed medical therapy for the preventive treatment of non-flow limiting vulnerable coronary lesions
  Interventions: Device: Sirolimus drug eluting ballooon therapy
- Guidelines-directed medical therapy (Active Comparator): Guidelines-directed medical therapy
  Interventions: Drug: Optimal guidelines-directed medical therapies (GDMT)

INTERVENTIONS:
Device: Sirolimus drug eluting ballooon therapy — Non-flow limiting vulnerable coronary plaques are treated using sirolimus drug eluting balloon therapy additional to guidelines directed medical therapy.
  Other Names: DEB-GDMT
  Arms: Sirolimus-eluting DEB (Selution SLR) therapy + Guidelines-directed medical therapy
Drug: Optimal guidelines-directed medical therapies (GDMT) — Optimal guidelines-directed medical therapies (GDMT) to reduce plaque burden and vulnerability for non-flow limiting vulnerable plaques
  Arms: Guidelines-directed medical therapy

SUMMARY:
The goal of this pilot clinical trial is to evaluate the use of the Selution SLR sirolimus-eluting balloon, in addition to guideline-directed medical therapy (GDMT), for the preventive treatment of non-flow-limiting vulnerable coronary lesions, compared to GDMT alone, in adult patients with multivessel coronary artery disease and a recent acute coronary syndrome (within 90 days).

The main research question is:

Does the use of the Selution SLR sirolimus-eluting balloon in combination with GDMT reduce the progression and vulnerability of non-flow-limiting vulnerable coronary plaques?

Participants will undergo

* PCI procedure with baseline IVUS-NIRS assessment
* Follow-up coronary angiography at 6 months with IVUS-NIRS assessment
* Clinical follow-up at 3, 6, and 24 months after study enrollment

ELIGIBILITY:
Inclusion Criteria:

Potential subjects must fulfill all following inclusion criteria:

1. Multivessel coronary artery disease with ACS within 90 days prior to inclusion and successful interventional treatment of the culprit lesion
2. Presence of ≥ 2 de novo non-culprit lesion without hemodynamic relevance in two different coronary vessels (demonstrated either by wire-based or angiography-based coronary physiology) and with MaxLCBI4mm ≥ 325 at baseline IVUS-NIRS
3. Age ≥ 18 years
4. Written informed consent

Exclusion Criteria:

Patients are not eligible if any of the following applies:

1. Non culprit lesion involving the left main and/or ostial left coronary artery, ostial left circumflex artery or ostial right coronary artery;
2. Non-culprit lesion in a previously stented segment (i.e. within 15 mm from the previously implanted stent);
3. Non-culprit lesion involving small vessel (<3.0 mm) deemed not suitable to PCI,
4. Non-culprit lesion located in a bypass graft or in a grafted vessel;
5. Severe renal impairment (eGFR<15ml/min/1.73m2) or patient on dialysis treatment;
6. Known pregnancy r breast-feeding patients;
7. Life expectancy <2 year due to other severe non-cardiac disease;
8. Legally incompetent to provide informed consent;
9. Partecipation in another clinical study with an investigational product

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Absolute change in the IVUS-NIRS derived lipid core burden index (MAXLCBI4mm) between baseline and 6-months follow-up. | Between baseline and 6-months follow-up.

SECONDARY OUTCOMES:
QCA parameter (minimal lumen diameter, MLD, mm) before and after intervention and at follow-up angiography. | pre procedure, immediately after the procedure and at 6(±30 days) months follow-up.
  Minimal lumen diameter (MLD, mm) before the intervention, immediately after the intervention and at follow up angiography.
QCA parameter (maximal diameter stenosis, MaxS,%) before and after intervention and at follow-up angiography. | pre procedure, immediately after the procedure and at 6(±30 days) months follow-up.
  Maximal diameter stenosis (MaxS,%) before the intervention, immediately after the intervention and at follow up angiography.
QCA parameter (reference vessel diameter, RVD, mm) before and after intervention and at follow-up angiography. | pre procedure, immediately after the procedure and at 6(±30 days) months follow-up.
  Reference vessel diameter (RVD, mm) before the intervention, immediately after the intervention and at follow up angiography.
QCA parameter (lesion lenght, LL, mm) before and after intervention and at follow-up angiography. | pre procedure, immediately after the procedure and at 6(±30 days) months follow-up.
  Lesion lenght (LL, mm) before the intervention, immediately after the intervention and at follow up angiography.
QFR parameters before and after the intervention and at follow-up angiography | pre procedure, immediately after the procedure and at 6(±30days) months follow-up.
  Quantitative Flow Ration (QFR) parameters before the intervention, immediately after the intervention and at follow-up angiography.
IVUS parameter (minimal lumen diameter, MLD, mm) before the intervention, immediately after the intervention and at follow-up angiography. | pre procedure, immediately after the procedure and at 6(±30days) months follow-up.
  Minimal lumen diameter (MLD, mm) before the intervention, immediately after the intervention and at follow-up angiography.
IVUS parameter (minimal lumen area, MLA, mm2) before the intervention, immediately after the intervention and at follow-up angiography. | pre procedure, immediately after the procedure and at 6(±30days) months follow-up.
  Minimal lumen area (MLA, mm2) before the intervention, immediately after the intervention and at follow-up angiography.
IVUS parameter (maximal diameter stenosis, MaxS,%) before the intervention, immediately after the intervention and at follow-up angiography. | pre procedure, immediately after the procedure and at 6(±30days) months follow-up.
  Maximal diameter stenosis (MaxS, %) before the intervention, immediately after the intervention and at follow-up angiography.
IVUS parameter (lumen volume, LV, mm3) before the intervention, immediately after the intervention and at follow-up angiography. | pre procedure, immediately after the procedure and at 6(±30days) months follow-up.
  Lumen volume (LV, mm3) before the intervention, immediately after the intervention and at follow-up angiography.
IVUS parameter (vessel volume, VV, mm3) before the intervention, immediately after the intervention and at follow-up angiography. | pre procedure, immediately after the procedure and at 6(±30days) months follow-up.
  Vessel volume (VV, mm3) before the intervention, immediately after the intervention and at follow-up angiography.
IVUS parameter (plaque burden, VV-LV) before the intervention, immediately after the intervention and at follow-up angiography. | pre procedure, immediately after the procedure and at 6(±30days) months follow-up.
  Plaque burden (VV-LV) before the intervention, immediately after the intervention and at follow-up angiography.
IVUS parameter (late lumen loss, LLL) before the intervention, immediately after the intervention and at follow-up angiography. | pre procedure, immediately after the procedure and at 6(±30days) months follow-up.
  Late lumen loss (LLL) before the intervention, immediately after the intervention and at follow-up angiography.
IVUS parameter (acute gain) before the intervention and immediately after the percutaneous intervention. | pre procedure and immediately after the procedure.
  Acute gain before the intervention (T0) and immediately after the percutaneous intervention (Tf).
IVUS parameter (disease progression) after the final result of index PCI (Tf) and at 6(±30days) month follow-up procedure. | immediately after the procedure and at 6(±30 days) months after the index PCI.
  Variation between the final result of index PCI (Tf) and procedure at 6(±30days) month follow-up (Tc).
Target Lesion Revascularization (TLR) | During hospitalization and at 6(±30days) month follow-up.
  Rate of target lesion revascularization (TLR) defined as urgent and non urgent
Target Vessel Revascularization (TVR) | During hospitalization and at 6(±30days) month follow-up.
  Rate of target vessel revascularization (TVR) defined as urgent and non-urgent.
Target Vessel Failure (TVF) | During hospitalization and at 6(±30days) month follow-up.
  Rate of target vessel failure, defined as cardiac death, target-vessel myocardial infarction and any target lesion revascularization.
Individual components of the composite target vessel failure (TVF) endpoint (defined as cardiac death, target-vessel myocardial infarction and any target lesion revascularization) | During hospitalization and at 6(±30days) month follow-up.
  Rate of the individual components of the composite target vessel failure (TVF) endpoint (defined as cardiac death, target-vessel myocardial infarction and any target lesion revascularization).
Major adverse cardiac events (MACE) defined as cardiac death, any myocardial infarction and any revascularization. | 6(± 30 days) months after the index PCI.
  Rate of major adverse cardiac events (MACE) defined as cardiac death, any myocardial infarction and any revascularization .
The individual components of the composite major adverse cardiac events (MACE- defined as cardiac death, any myocardial infarction and any revascularization). | 6(± 30 days) months after the index PCI.
  Rate of the individual components of the composite MACE endpoint (defined as cardiac death, any myocardial infarction, any revascularization).
Stroke | 6(± 30 days) months after the index PCI.
  Rate of stroke.

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Cardiocentro Ticino - EOC, Lugano, Switzerland

IPD SHARING:
Plan to Share IPD: No
The final study data will be disseminated to the scientific community through the publication of results in peer-reviewed journals, ensuring accessibility to researchers and healthcare professionals.